CLINICAL TRIAL: NCT04997980
Title: aMsa and amiOdarone Study in cArdiaC Arrest
Acronym: MOSAIC
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other); Oslo University Hospital (Other); The Hospital of Vestfold (Other)
Responsible Party: Principal Investigator, Simone Savastano, principal investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: IRCCSPSM 1
Record Dates: First submitted 2021-07-18; First posted 2021-08-10 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: AMSA; amiodarone; Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Amiodarone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amiodarone group: Patients who did receive amiodarone during the attempt of resuscitation
  Interventions: Drug: Amiodarone Injection
- NO Amiodarone: Patients who did receive amiodarone during the attempt of resuscitation

INTERVENTIONS:
Drug: Amiodarone Injection
  Groups: Amiodarone group

SUMMARY:
Investigators' aim is to assess whether the administration of amiodarone during resuscitation could cause a reduction of the values of the amplitude spectral area (AMSA).

Amiodarone is recommended for the treatment of cardiac arrest due to ventricular tachycardia/ventricular fibrillation (VT/VF) ( with a low level of recommendation cause of conflicting results. AMSA is a parameter expressing the amplitude of VF and it has been shown to predict defibrillation success and the return of spontaneous circulation (ROSC). No data are available so far about the impact of amiodarone administration on AMSA values.

DETAILED DESCRIPTION:
The primary study endpoint of the present study is to determine whether patients who received amiodarone during advanced resuscitation had lower values of AMSA as compared to those who did not receive amiodarone.

Secondary endpoints

The secondary endpoints of this study are:

1. To assess, after correction for confounders, the rate of successful defibrillation, the rate of ROSC and the rate of short-term survival (survived event or survival to hospital discharge according to the available data) both in the amiodarone and non-amiodarone group.
2. To assess the role of AMSA for shock success and ROSC prediction in amiodarone group and in non-amiodarone group.

Type of study. This is a multicentre study based on a retrospective analysis of prospectically collected data.

Study population All the out-of-hospital cardiac arrests (OHCA) which occurred from January 1st, 2015 to December 31st, 2020 will be considered for the present study. In the analysis the investigators will include only those patients who received at least one shock for ventricular fibrillation during advanced resuscitation regardless whether or not the presenting rhythm was shockable or non-shockable.

The study cohort will involve cases retrieved from the Lombardia CARe registry (Lombardia Cardiac Arrest Registry NCT03197142), from the registry of Oslo and Vestfold

Data Collection Data from different databases will be integrated and combined in a single ad hoc database for statistical analysis.

For every shock, both pre-shock carbon dioxide at the end ot the tidal volume (ETCO2) and pre-shock AMSA will be calculated. The median ETCO2 value in the minute before the shock (METCO2) will be computed automatically either from a capnogram, when available, applying the algorithm described by Aramendi et al, or from the defibrillator with a ETCO2 monitoring feature. AMSA will be computed using a 2-second-pre-shock ECG interval, free of chest compression artifacts, leaving a 1-second guard before the shock. The electrocardiogram (ECG) will be bandpass filtered (0.5-30Hz) and the fast Fourier transform computed to obtain AMSA in the 2-48 Hz bandwidth.

For each patient all the pre-hospital variables will be included according to the 2014 Utstein recommendations and the number of shocks will be computed. The mean value of both ETCO2 and of AMSA will be calculated.

Statistical analysis Categorical variables will be compared with the Chi-square test and presented as number and percentage. Continuous variables will be compared with the t-test and presented as mean ± standard deviation, or compared with the Mann-Whitney test and presented as median and interquartile range (IQR) according to normal distribution tested with the D'Agostino-Pearson test. A multivariable regression model will be fitted both for shock success and for ROSC (including all non-correlated potential predictors) and to test the effect of amiodarone on AMSA values after correction for confounders.

The values of AMSA in the amiodarone and in the non-amiodarone group will then be compared in two groups of shocks randomly matched and identified via propensity score matching, so that they are homogeneous for time to shock, pre-shock ETCO2, outcome of defibrillation and the age of the patients.

ELIGIBILITY:
Inclusion Criteria:

clinical:

* patients with out-of-hospital cardiac arrest
* shockable presenting rhythm
* resuscitation attempted
* advanced resuscitation attempted

technical: - VF cardiac arrest (and not VT)

Exclusion Criteria:

clinical:

* non-shockable presenting rhythm
* resuscitation not attempted

technical:

- AMSA not evaluable

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the consecutive patients suffering of out-of-hospital cardiac arrest with a shockable presenting rhythm and receiving an advanced attempt of resuscitation.
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
AMSA values | through study completion, an average of 1 year
  to determine whether AMSA values in the Amiodarone group are lower than in the NO Amiodarone gorup

SECONDARY OUTCOMES:
Successful defibrilaltion | through study completion, an average of 1 year
  to assess the rate of successful defibrillation in the Amiodarone and in the NO Amiodarone group
ROSC | through study completion, an average of 1 year
  to assess the rate of ROSC in the Amiodarone and in the NO Amiodarone group
Survived event | through study completion, an average of 1 year
  to assess the rate of "survived event" in the Amiodarone and in the NO Amiodarone group
Survival to hospital discharge | through study completion, an average of 1 year
  to assess the rate of survival to hospital discharge in the Amiodarone and in the NO Amiodarone group
Prediction | through study completion, an average of 1 year
  to verify if AMSA maintain its predictive role for defibrillation success and ROSC also in the Amiodarone group

CONTACTS AND LOCATIONS:
Locations (4):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- Norway (2):
  - Oslo University Hospital, Oslo
  - Vestfold Hospital trust, Tønsberg
- BioRes Research Group, Bilbao, Spain

IPD SHARING:
Plan to Share IPD: No
Data could be shared under motivated request following a proposal.

REFERENCES:
- [Background] Schwartz PJ, Zaza A. The Sicilian Gambit revisited--theory and practice. Eur Heart J. 1992 Nov;13 Suppl F:23-9. doi: 10.1093/eurheartj/13.suppl_f.23. No abstract available. PMID 1478220
- [Background] Zipes DP, Prystowsky EN, Heger JJ. Amiodarone: electrophysiologic actions, pharmacokinetics and clinical effects. J Am Coll Cardiol. 1984 Apr;3(4):1059-71. doi: 10.1016/s0735-1097(84)80367-8. PMID 6368644
- [Background] Marinchak RA, Friehling TD, Kline RA, Stohler J, Kowey PR. Effect of antiarrhythmic drugs on defibrillation threshold: case report of an adverse effect of mexiletine and review of the literature. Pacing Clin Electrophysiol. 1988 Jan;11(1):7-12. doi: 10.1111/j.1540-8159.1988.tb03925.x. PMID 2449675
- [Background] Zhou L, Chen BP, Kluger J, Fan C, Chow MS. Effects of amiodarone and its active metabolite desethylamiodarone on the ventricular defibrillation threshold. J Am Coll Cardiol. 1998 Jun;31(7):1672-8. doi: 10.1016/s0735-1097(98)00160-0. PMID 9626850
- [Background] Hohnloser SH, Dorian P, Roberts R, Gent M, Israel CW, Fain E, Champagne J, Connolly SJ. Effect of amiodarone and sotalol on ventricular defibrillation threshold: the optimal pharmacological therapy in cardioverter defibrillator patients (OPTIC) trial. Circulation. 2006 Jul 11;114(2):104-9. doi: 10.1161/CIRCULATIONAHA.106.618421. Epub 2006 Jul 3. PMID 16818810
- [Background] Jung W, Manz M, Pizzulli L, Pfeiffer D, Luderitz B. Effects of chronic amiodarone therapy on defibrillation threshold. Am J Cardiol. 1992 Oct 15;70(11):1023-7. doi: 10.1016/0002-9149(92)90354-2. PMID 1414899
- [Background] Fain ES, Lee JT, Winkle RA. Effects of acute intravenous and chronic oral amiodarone on defibrillation energy requirements. Am Heart J. 1987 Jul;114(1 Pt 1):8-17. doi: 10.1016/0002-8703(87)90300-0. PMID 3604876
- [Background] Soar J, Berg KM, Andersen LW, Bottiger BW, Cacciola S, Callaway CW, Couper K, Cronberg T, D'Arrigo S, Deakin CD, Donnino MW, Drennan IR, Granfeldt A, Hoedemaekers CWE, Holmberg MJ, Hsu CH, Kamps M, Musiol S, Nation KJ, Neumar RW, Nicholson T, O'Neil BJ, Otto Q, de Paiva EF, Parr MJA, Reynolds JC, Sandroni C, Scholefield BR, Skrifvars MB, Wang TL, Wetsch WA, Yeung J, Morley PT, Morrison LJ, Welsford M, Hazinski MF, Nolan JP; Adult Advanced Life Support Collaborators. Adult Advanced Life Support: 2020 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science with Treatment Recommendations. Resuscitation. 2020 Nov;156:A80-A119. doi: 10.1016/j.resuscitation.2020.09.012. Epub 2020 Oct 21. PMID 33099419
- [Background] Sanfilippo F, Corredor C, Santonocito C, Panarello G, Arcadipane A, Ristagno G, Pellis T. Amiodarone or lidocaine for cardiac arrest: A systematic review and meta-analysis. Resuscitation. 2016 Oct;107:31-7. doi: 10.1016/j.resuscitation.2016.07.235. Epub 2016 Aug 3. PMID 27496262
- [Background] Tagami T, Yasunaga H, Yokota H. Antiarrhythmic drugs for out-of-hospital cardiac arrest with refractory ventricular fibrillation. Crit Care. 2017 Mar 21;21(1):59. doi: 10.1186/s13054-017-1639-8. PMID 28320450
- [Background] Tagami T, Matsui H, Tanaka C, Kaneko J, Kuno M, Ishinokami S, Unemoto K, Fushimi K, Yasunaga H. Amiodarone Compared with Lidocaine for Out-Of-Hospital Cardiac Arrest with Refractory Ventricular Fibrillation on Hospital Arrival: a Nationwide Database Study. Cardiovasc Drugs Ther. 2016 Oct;30(5):485-491. doi: 10.1007/s10557-016-6689-7. PMID 27618826
- [Background] Chowdhury A, Fernandes B, Melhuish TM, White LD. Antiarrhythmics in Cardiac Arrest: A Systematic Review and Meta-Analysis. Heart Lung Circ. 2018 Mar;27(3):280-290. doi: 10.1016/j.hlc.2017.07.004. Epub 2017 Aug 23. PMID 28988724
- [Background] Zhao H, Fan K, Feng G. Amiodarone and/or lidocaine for cardiac arrest: A Bayesian network meta-analysis. Am J Emerg Med. 2020 Oct;38(10):2185-2193. doi: 10.1016/j.ajem.2020.06.074. Epub 2020 Jul 5. PMID 33071078
- [Background] Ong ME, Pellis T, Link MS. The use of antiarrhythmic drugs for adult cardiac arrest: a systematic review. Resuscitation. 2011 Jun;82(6):665-70. doi: 10.1016/j.resuscitation.2011.02.033. Epub 2011 Mar 27. PMID 21444143
- [Background] Kudenchuk PJ, Leroux BG, Daya M, Rea T, Vaillancourt C, Morrison LJ, Callaway CW, Christenson J, Ornato JP, Dunford JV, Wittwer L, Weisfeldt ML, Aufderheide TP, Vilke GM, Idris AH, Stiell IG, Colella MR, Kayea T, Egan D, Desvigne-Nickens P, Gray P, Gray R, Straight R, Dorian P; Resuscitation Outcomes Consortium Investigators. Antiarrhythmic Drugs for Nonshockable-Turned-Shockable Out-of-Hospital Cardiac Arrest: The ALPS Study (Amiodarone, Lidocaine, or Placebo). Circulation. 2017 Nov 28;136(22):2119-2131. doi: 10.1161/CIRCULATIONAHA.117.028624. Epub 2017 Sep 13. PMID 28904070
- [Background] Kudenchuk PJ, Cobb LA, Copass MK, Cummins RO, Doherty AM, Fahrenbruch CE, Hallstrom AP, Murray WA, Olsufka M, Walsh T. Amiodarone for resuscitation after out-of-hospital cardiac arrest due to ventricular fibrillation. N Engl J Med. 1999 Sep 16;341(12):871-8. doi: 10.1056/NEJM199909163411203. PMID 10486418
- [Background] Dorian P, Cass D, Schwartz B, Cooper R, Gelaznikas R, Barr A. Amiodarone as compared with lidocaine for shock-resistant ventricular fibrillation. N Engl J Med. 2002 Mar 21;346(12):884-90. doi: 10.1056/NEJMoa013029. PMID 11907287
- [Background] Ristagno G, Li Y, Fumagalli F, Finzi A, Quan W. Amplitude spectrum area to guide resuscitation-a retrospective analysis during out-of-hospital cardiopulmonary resuscitation in 609 patients with ventricular fibrillation cardiac arrest. Resuscitation. 2013 Dec;84(12):1697-703. doi: 10.1016/j.resuscitation.2013.08.017. Epub 2013 Sep 1. PMID 24005007
- [Background] Ristagno G, Mauri T, Cesana G, Li Y, Finzi A, Fumagalli F, Rossi G, Grieco N, Migliori M, Andreassi A, Latini R, Fornari C, Pesenti A; Azienda Regionale Emergenza Urgenza Research Group. Amplitude spectrum area to guide defibrillation: a validation on 1617 patients with ventricular fibrillation. Circulation. 2015 Feb 3;131(5):478-87. doi: 10.1161/CIRCULATIONAHA.114.010989. Epub 2014 Dec 2. PMID 25466976
- [Background] Salcido DD, Schmicker RH, Kime N, Buick JE, Cheskes S, Grunau B, Zellner S, Zive D, Aufderheide TP, Koller AC, Herren H, Nuttall J, Sundermann ML, Menegazzi JJ; Resuscitation Outcomes Consortium Investigators. Effects of intra-resuscitation antiarrhythmic administration on rearrest occurrence and intra-resuscitation ECG characteristics in the ROC ALPS trial. Resuscitation. 2018 Aug;129:6-12. doi: 10.1016/j.resuscitation.2018.05.028. Epub 2018 May 24. PMID 29803703
- [Background] Frigerio L, Baldi E, Aramendi E, Chicote B, Irusta U, Contri E, Palo A, Compagnoni S, Fracchia R, Iotti G, Oltrona Visconti L, Savastano S; Lombardia CARe Researchers. End-tidal carbon dioxide (ETCO2) and ventricular fibrillation amplitude spectral area (AMSA) for shock outcome prediction in out-of-hospital cardiac arrest. Are they two sides of the same coin? Resuscitation. 2021 Mar;160:142-149. doi: 10.1016/j.resuscitation.2020.10.032. Epub 2020 Nov 10. PMID 33181229
- [Background] Ristagno G, Gullo A, Berlot G, Lucangelo U, Geheb E, Bisera J. Prediction of successful defibrillation in human victims of out-of-hospital cardiac arrest: a retrospective electrocardiographic analysis. Anaesth Intensive Care. 2008 Jan;36(1):46-50. doi: 10.1177/0310057X0803600108. PMID 18326131
- [Background] Aiello S, Perez M, Cogan C, Baetiong A, Miller SA, Radhakrishnan J, Kaufman CL, Gazmuri RJ. Real-Time Ventricular Fibrillation Amplitude-Spectral Area Analysis to Guide Timing of Shock Delivery Improves Defibrillation Efficacy During Cardiopulmonary Resuscitation in Swine. J Am Heart Assoc. 2017 Nov 4;6(11):e006749. doi: 10.1161/JAHA.117.006749. PMID 29102980
- [Background] Hulleman M, Salcido DD, Menegazzi JJ, Souverein PC, Tan HL, Blom MT, Koster RW. Predictive value of amplitude spectrum area of ventricular fibrillation waveform in patients with acute or previous myocardial infarction in out-of-hospital cardiac arrest. Resuscitation. 2017 Nov;120:125-131. doi: 10.1016/j.resuscitation.2017.08.219. Epub 2017 Aug 24. PMID 28844935
- [Background] Ruggeri L, Semeraro F, Ristagno G. Amplitude spectrum area: The "clairvoyance" during resuscitation in the era of predictive medicine. Resuscitation. 2017 Nov;120:A5-A6. doi: 10.1016/j.resuscitation.2017.09.011. Epub 2017 Sep 18. No abstract available. PMID 28928017
- [Background] Hulleman M, Salcido DD, Menegazzi JJ, Souverein PC, Tan HL, Blom MT, Koster RW. Ventricular fibrillation waveform characteristics in out-of-hospital cardiac arrest and cardiovascular medication use. Resuscitation. 2020 Jun;151:173-180. doi: 10.1016/j.resuscitation.2020.02.027. Epub 2020 Mar 10. PMID 32169604
- [Background] Aramendi E, Elola A, Alonso E, Irusta U, Daya M, Russell JK, Hubner P, Sterz F. Feasibility of the capnogram to monitor ventilation rate during cardiopulmonary resuscitation. Resuscitation. 2017 Jan;110:162-168. doi: 10.1016/j.resuscitation.2016.08.033. Epub 2016 Sep 23. PMID 27670357
- [Background] Freedman MD, Somberg JC. Pharmacology and pharmacokinetics of amiodarone. J Clin Pharmacol. 1991 Nov;31(11):1061-9. doi: 10.1002/j.1552-4604.1991.tb03673.x. PMID 1753010